CLINICAL TRIAL: NCT05654909
Title: Prehospital Assessment Units - a Matched Cohort Study
Status: Completed | Type: Observational
Sponsor: Prehospital Center, Region Zealand (Other)
Responsible Party: Principal Investigator, Signe Amalie Wolthers, MD, Prehospital Center, Region Zealand
Other Study IDs: PHV_2022
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-02-16 (Actual); Status verified 2023-02

CONDITIONS: Pneumonia; Urinary Tract Infections; Fall; Infections; GI Disorders; Orthopedic Disorder
MeSH Terms: conditions — Pneumonia; Urinary Tract Infections; Infections; Digestive System Diseases; Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PAU group: The PAU group were patients calling 1-1-2 assigned for the prehospital assessment unit,
  Interventions: Procedure: Prehospital assessment unit
- non PAU group: The non PAU group were selected from the 1-1-2 calls (the European version of 9-1-1) EMS and were collected based on the same criteria as the patients assessed by the PAU. The control ratio was 1:10 for cases to increase power. Controls were matched on sex and age (within 5-year ranges). Matching was performed using incidence density sampling, where controls were selected for each case on the week of 1-1-2 call.

INTERVENTIONS:
Procedure: Prehospital assessment unit — The prehospital assessment unit was developed to provide a paramedic responding by car to 1-1-2 calls in the area of Region Zealand. Further details are mentioned in the description.
  Groups: PAU group

SUMMARY:
This study aimed to evaluate the prehospital assessment unit (PAU) by admission within 48 hours, 7 days, respectively and on survival.

The PAU should increase focus on a patient-centered approach with the capability to make advanced assessments of patients to reduce unnecessary transportation. Further, this paramedic assessment program could positively impact the healthcare system by reducing admissions to emergency departments.

The PAU is operated by paramedics who have additional education, and they are capable of testing and monitoring certain conditions at the scene - in the home of the patients. The paramedics decide if the patient requires admission to the hospital or if the patient could stay at home. They are consulting physicians on call by phone.

This retrospective cohort study included data from patients assessed by the PAU between November 1st 2021, and October 1st 2022.

Non-PAU patients were selected from the 1-1-2 calls (the European version of 9-1-1) EMS and were collected based on the same criteria as the patients assessed by the PAU. The control ratio was 1:10 for cases to increase power. The non-PAU patients were matched on sex and age (within 5-year ranges). Matching was performed using incidence density sampling, where controls were selected for each case on the week of 1-1-2 call.

DETAILED DESCRIPTION:
The demand for healthcare is increasing, stressing the need for adaptive Emergency Medical Services (EMS). This development was also illustrated in a Danish cohort study from 2017. The authors reported an increase in the annual number of patients assessed by EMS by 67% between 2007 and 2014.Thus, the traditional role of paramedics is changing to establish a bridge between the community and the hospital by offering primary care services. Paramedic assessment units (PAU) were implemented in Region Zealand, Denmark in 2021 to accommodate the increased demand. The PAU should increase focus on a patient-centered approach with the capability to make advanced assessments of patients to reduce unnecessary transportation. Further, this paramedic assessment program could positively impact the healthcare system by reducing admissions to emergency departments.

While this approach is new in Denmark, variations of the approach have been implemented internationally for more than two decades.The PAU can be compared with the community paramedic units. Different community paramedic programs have arisen to address the regional requirements; different regional and national operation environments explain this regarding the population density and level of healthcare service. No exact definition is present, but these assessment programs generally focus on frail elderly and other high-needs patients.

The PAU is operated by paramedics who have additional education, and they do have point-of-care test facilities (POCT). The paramedics can monitor saturation, blood pressure and electrocardiogram, all of which are standard equipment of ambulances in Region Zealand. Further, the paramedic can measure C-reactive protein, analyse urine test strips (pH, glucose, acetoacetate, leucocytes, nitrite, protein and erythrocytes), blood glucose and analyse blood gas (pH, pO2, pCO2, lactate, sodium, potassium, calcium and creatinine).

The patients assessed by the PAU had four possible destinations: admittance to the E-Hospital, a unique regional arrangement in which the patient stays at home but is under virtual surveillance by physicians and nurses. Alternatively, the patient was admitted to the E-hospital at local acute community-based facilities. Third, the patient was admitted to the emergency department at the hospital and finally, the PAU examined the patient at home without further follow-up. The decision was made between the physicians at the E-Hospital and the paramedic on the scene.

While the evidence supporting PAU is promising, convincing data from well-designed studies focusing on the impact of PAU on health outcomes and patient safety are still being determined.

This retrospective cohort study was conducted to compare individuals treated by PAU with a control group of matched individuals not treated by PAU. Thus, the primary objective of this study was:

* To identify patients among cases who were admitted to the emergency department within 48 hours and 7 days after consultation with the PAU, respectively.
* Secondary, to identify patients admitted to the emergency department within 6 hours from the initial call to the medical emergency number.
* Finally, to identify 30-day survival.

ELIGIBILITY:
Inclusion Criteria:

* expectations of undergoing an uncomplicated illness progression
* green or yellow level of triage based on the ABCDE approach (red, orange, yellow, green, blue levels of triage.

Exclusion Criteria:

* gynaecological disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients in the Region Zealand calling 1-1-2 during the study period
Sampling Method: Non-Probability Sample
Enrollment: 10849 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2023-01-01 (Actual)

PRIMARY OUTCOMES:
Admission within 48 hours | 48 hours
  Dichotomous variable of admission within two days after intial call
Admission within 7 days | 7 dats
  Dichotomous variable of admission within seven days after intial call

SECONDARY OUTCOMES:
Admission within 6 hours | 6 hours
  Dichotomous variable of admission within 6 hours from intial call
30-day survival | 30-day
  30-day survival from initial call

CONTACTS AND LOCATIONS:
Locations (1):
- Prehospital Center, Næstved, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Andersen MS, Johnsen SP, Sorensen JN, Jepsen SB, Hansen JB, Christensen EF. Implementing a nationwide criteria-based emergency medical dispatch system: a register-based follow-up study. Scand J Trauma Resusc Emerg Med. 2013 Jul 9;21:53. doi: 10.1186/1757-7241-21-53. PMID 23835246
- [Background] Christensen EF, Bendtsen MD, Larsen TM, Jensen FB, Lindskou TA, Holdgaard HO, Hansen PA, Johnsen SP, Christiansen CF. Trends in diagnostic patterns and mortality in emergency ambulance service patients in 2007-2014: a population-based cohort study from the North Denmark Region. BMJ Open. 2017 Aug 21;7(8):e014508. doi: 10.1136/bmjopen-2016-014508. PMID 28827233
- [Derived] Wolthers SA, Blomberg SNF, Breindahl N, Anjum S, Hagi-Pedersen D, Ersboll A, Andersen LB, Christensen HC. Association between using a prehospital assessment unit and hospital admission and mortality: a matched cohort study. BMJ Open. 2023 Sep 22;13(9):e075592. doi: 10.1136/bmjopen-2023-075592. PMID 37739475